CLINICAL TRIAL: NCT00585247
Title: Combining Topical Imiquimod 5% Cream With a Pulsed Dye Laser to Treat Port Wine Stain Birthmarks
Acronym: Aldara
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Kristen Kelly, M.D., Professor Departments of Dermatology and Surgery, University of California, Irvine
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 20064815
Record Dates: First submitted 2007-12-18; First posted 2008-01-03 (Estimated); Results first posted 2018-04-04 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Port Wine Stain
Keywords: birthmarks
MeSH Terms: conditions — Port-Wine Stain | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Imiquimod (Experimental): Combining Topical Imiquimod 5% Cream With a Pulsed Dye Laser to Treat Port Wine Stain Birthmarks
  Interventions: Drug: Imiquimod
- Placebo (Placebo Comparator): Combining Topical Imiquimod 5% Cream With a Pulsed Dye Laser to Treat Port Wine Stain Birthmarks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Imiquimod — Combining Topical Imiquimod 5% Cream With a Pulsed Dye Laser to Treat Port Wine Stain Birthmarks
  Other Names: Combining Topical Imiquimod 5% Cream With a Pulsed Dye Laser
  Arms: Imiquimod
Other: Placebo — Combining Topical Imiquimod 5% Cream With a Pulsed Dye Laser to Treat Port Wine Stain Birthmarks
  Other Names: Combining Topical Imiquimod 5% Cream With a Pulsed Dye Laser
  Arms: Placebo

SUMMARY:
Port wine stains are red birthmarks that without treatment persist for a lifetime. They are frequently found on the face and can be conspicuous and disfiguring, negatively impacting social interactions for these patients. Treating Port wine stains is difficult. The standard of care is to use laser treatment, but over 80% of patients fail to completely clear despite multiple treatments. The growth of additional blood vessels (angiogenesis) following the Laser treatment is likely an important factor in why these lesions persist despite therapy.

DETAILED DESCRIPTION:
Imiquimod is a topical cream that affects the immune response and has been noted to inhibit blood vessel formation. It has been used to successfully treat other vascular growths such as hemangiomas. The research can use imiquimod cream 5% cream apply to port wine stains after laser therapy to improve lightening of port wine stains. The imiquimod 5% cream cream apply to Port wine stains everyday for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Port Wine Stain birthmark
* Male and female subjects of any age who are in good health.
* Fitzpatrick skin type I-VI

Exclusion Criteria:

* Pregnant or lactating
* History of cutaneous photosensitivity
* History of hypersensitivity to imiquimod 5% cream or any of its components
* History of photodermatoses

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen M Kelly, M.D, Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (1):
- Beckman Laser Institute Medical and Surgical Cilnic, Irvine, California, United States

REFERENCES:
- [Result] Tremaine AM, Armstrong J, Huang YC, Elkeeb L, Ortiz A, Harris R, Choi B, Kelly KM. Enhanced port-wine stain lightening achieved with combined treatment of selective photothermolysis and imiquimod. J Am Acad Dermatol. 2012 Apr;66(4):634-41. doi: 10.1016/j.jaad.2011.11.958. Epub 2012 Jan 14. PMID 22244840
- See also: Enhanced port-wine stain lightening achieved with combined treatment of selective photothermolysis and imiquimod — http://www.ncbi.nlm.nih.gov/pubmed/22244840

RESULTS

PARTICIPANT FLOW:
Groups:
- Imiquimod: Combining Topical Imiquimod 5% Cream With a Pulsed Dye Laser to Treat Port Wine Stain Birthmarks
  Imiquimod: Combining Topical Imiquimod 5% Cream With a Pulsed Dye Laser to Treat Port Wine Stain Birthmarks
  Healthy individuals with PWS (n = 14) were treated with PDL and then randomized to apply post treatment Imiquimod 5% cream for 8 weeks for 57 PWS sites (multiple sites per patient)
- Placebo: Combining Topical Imiquimod 5% Cream With a Pulsed Dye Laser to Treat Port Wine Stain Birthmarks
  Placebo: Combining Topical Imiquimod 5% Cream With a Pulsed Dye Laser to Treat Port Wine Stain Birthmarks
  Healthy individuals with PWS (n = 13) were treated with PDL and then randomized to apply post treatment placebo cream for 8 weeks for 57 PWS sites (multiple sites per patient)
Period: Overall Study
Arm/Group | Imiquimod | Placebo
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 27 subjects was enrolled to the study for 57 PWS sites (multiple sites per patient).
Groups:
- Imiquimod: Combining Topical Imiquimod 5% Cream With a Pulsed Dye Laser to Treat Port Wine Stain Birthmarks
  Imiquimod: Combining Topical Imiquimod 5% Cream With a Pulsed Dye Laser to Treat Port Wine Stain Birthmarks were treated with PDL and then randomized to apply post treatment imiquimod 5% cream for 8 weeks.
- Placebo: Combining Topical Imiquimod 5% Cream With a Pulsed Dye Laser to Treat Port Wine Stain Birthmarks
  Placebo: Combining Topical Imiquimod 5% Cream With a Pulsed Dye Laser to Treat Port Wine Stain Birthmarks were treated with PDL and then randomized to apply post treatment placebo cream for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Imiquimod | Placebo | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 0 | 4
  Between 18 and 65 years | 9 | 13 | 22
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: Participants]
  United States | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in a* and E at 8 Weeks
Description: Change in a* and ΔE is a way to quantify PWS treatment outcome: a* is the erythema of the vascular lesions and varies from +60 for green to -60 for red with a value of +9.28 for Normal Skin. Higher a* values indicates a greater reduction in erythema hence better treatment outcome. ΔE detects all three dimensions of colorspace (L*a*b*) and represents the difference in color between normal and PWS skin. Range of ΔE is 0 to 100. Higher values indicates improved treatment efficacy by greater skin color improvement.
Time Frame: 8 weeks baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Imiquimod | Placebo
Number analyzed (Participants) | 14 | 13
units on a scale
  a* | 1.27 (1.76) | 0.43 (1.63)
  ΔE | 4.08 (3.39) | 2.59 (1.54)

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- Imiquimod: Combining Topical Imiquimod 5% Cream With a Pulsed Dye Laser to Treat Port Wine Stain Birthmarks
  Imiquimod: Combining Topical Imiquimod 5% Cream With a Pulsed Dye Laser to Treat Port Wine Stain Birthmarks
  Healthy individuals with PWS (n = 24) were treated with PDL and then randomized to apply post treatment Imiquimod 5% cream for 8 weeks for 57 PWS sites (multiple sites per patient)
- Placebo: Combining Topical Imiquimod 5% Cream With a Pulsed Dye Laser to Treat Port Wine Stain Birthmarks
  Placebo: Combining Topical Imiquimod 5% Cream With a Pulsed Dye Laser to Treat Port Wine Stain Birthmarks
  Healthy individuals with PWS (n = 24) were treated with PDL and then randomized to apply post treatment placebo cream for 8 weeks for 57 PWS sites (multiple sites per patient)
Arm/Group | Imiquimod | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13

LIMITATIONS AND CAVEATS:
Effects were evaluated after a single treatment and duration of effect is unknown

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No